CLINICAL TRIAL: NCT06370910
Title: Comparison of Low-Level Laser Therapy With Cryotherapy in Postpartum Women With Laceration and/or Episiotomy on Perineal and Vulvar Pain Reduction
Brief Title: Comparison Low-Level Laser Therapy With Cryotherapy in Parturients With Laceration and/or Episiotomy on Pain Reduction
Acronym: CL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Elen Cristine Boniatti Constant, Investigador Principal, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 58569421.5.0000.5327
Record Dates: First submitted 2024-04-01; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Episiotomy; Complications; Laceration
Keywords: Cryotherapy; Low level Laser Therapy;
MeSH Terms: conditions — Lacerations | interventions — Low-Level Light Therapy; Cryotherapy

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Active Comparator): Cryotherapy will be performed using a glove containing crushed ice applied to the perineum region for 20 minutes, starting within 12 hours postpartum. The patients will be evaluated before the application, immediately after the application, immediately after the application and in 24 hours after the application.
  A glove containing crushed ice will be used because it is more anatomical and extends throughout the perineum region. The indicates that ice on the surface has the ability to decrease the temperature of the skin and intramuscular tissue. Compared to other cryotherapy techniques like gel and frozen pea pack, ice pack is the most adopted technique for perineal pain relief.
  The application time depends on the study, which indicates that 20 minutes is enough time to cause a reduction and relief of pain in the participants of their study.
  Interventions: Other: Low-Level Laser Therapy
- Low-Level Laser Therapy (Active Comparator): Within 12 hours postpartum, red light radiation will be applied at the site of the injury, with 3 joules applied promptly. The non-contact technique will be used, maintaining a distance of 2 cm between each point. Subsequently, infrared laser will be applied using conventional contact technique, around the extent of the injury. 6 joules will be applied punctually, also with a distance of 2 cm between each point. The LLLT device used will be the DMC brand Therapy EC, portable, with a lithium-ion battery. The red laser will have a wavelength of 660nm (+- 10 nm), with an emitter power of 100 mw (+- 20%). The infrared laser will have a wavelength of 808 nm (+- 10), with an emitter power of 100 mw (+- 20%).
  Interventions: Other: Low-Level Laser Therapy

INTERVENTIONS:
Other: Low-Level Laser Therapy — The patient will be submitted to evaluation through a questionnaire, which will be the patient's evaluation form, which will be elaborated by the researcher (Appendix A). Next, pain and edema will be evaluated, using the VAS scales, Mc Gill scale and REEDA scale, after this process, the therapy will be applied, and the patient will be randomly selected for cryotherapy or LLLT. After application, the patient will be evaluated immediately and the scales applied again and after 24 hours.
  Other Names: Cryotherapy

SUMMARY:
The changes that occur during pregnancy can lead to symptoms and complaints for women. Vaginal delivery has several benefits for both the mother and baby; however, during labor, some injuries may occur, such as lacerations and episiotomies. It is known that the postpartum period is when the body is involuting to its pre-pregnancy state. The perineal pain caused by these injuries during childbirth is a determining factor for recovery, and it may affect not only the physical but also the psychological well-being of women. Therefore, it is necessary to employ techniques that can alleviate pain and edema in the immediate postpartum period, directly influencing recovery.

Objective: To compare the use of photobiomodulation with cryotherapy in the immediate postpartum period of 2 hours in parturients who suffered 1st and 2nd-degree lacerations and/or episiotomies.

Methods: A randomized clinical trial will be conducted to compare two interventions. Data collection will be through a questionnaire and scales for the evaluation of pain and edema, with women who experienced vaginal delivery and those who suffered 1st and 2nd-degree lacerations or episiotomies.

Expected results: Reduction of pain, edema, and inflammatory processes with non-pharmacological techniques, leading to greater comfort and better postpartum recovery.

DETAILED DESCRIPTION:
Faced with the scarcity of evidence indicating the best approach to reducing edema and relieving pain in the postpartum period, there is a need to evaluate new methods for pain relief during this time to ensure better well-being for women in the postpartum period.

Lacerations and episiotomies, which can occur during vaginal delivery, exacerbate this pain, making it even more necessary to utilize resources to alleviate discomfort and perineal and vulvar edema, which can consequently worsen pain.

The postpartum period is challenging, with numerous adjustments, and pain can be debilitating, making this period particularly challenging. However, it is possible to minimize it with non-pharmacological interventions.

Cryotherapy has proven to be a valuable resource already utilized in the immediate postpartum period, and low-intensity laser therapy has also demonstrated effectiveness in pain relief, both with low associated risks and costs.

Therefore, it is crucial to compare which therapeutic approach is most effective during the immediate postpartum period.

While vaginal delivery offers many benefits, such as rapid recovery, it can be associated with perineal trauma, leading to pain, breastfeeding difficulties, and discomfort, which directly interfere with activities of daily living The use of an ice pack is inexpensive and effective in relieving pain in the immediate postpartum period, whereas low-level laser therapy (LLLT) promotes tissue repair, enhances wound healing, reduces inflammatory responses, and alleviates pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who underwent vaginal delivery;
2. Had a grade 1 or grade 2 laceration;
3. Have undergone episiotomy;

Exclusion Criteria:

1. Patient who underwent cesarean section;
2. With Help Syndrome;
3. They presented immediate postpartum hemorrhage;
4. They had unstable vital signs in the immediate postpartum period;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
To compare two techniques: Low-level laser and cryotherapy | 24 horas
  The use of low-level laser therapy or cryotherapy to alleviate pain. Cryotherapy was performed using a glove containing crushed ice, applied to the perineal region for 20 minutes, initiated within 12 hours postpartum. Patients were evaluated before the application, immediately after the application, and 24 hours after the application. Low-level laser therapy, as well as cryotherapy, was applied within 12 hours after delivery, targeting the site of the injury with red radiation. The applied dose was 3 joules, administered in a punctual manner, using a non-contact technique, with a distance of 2 cm between each point. Subsequently, infrared laser therapy was applied using conventional contact technique around the extent of the injury, with a punctual application of 6 joules, also maintaining a distance of 2 cm between each point.

SECONDARY OUTCOMES:
Pain reduction assessed by the Visual Analog Scale (VAS). | 24 hours
  The Visual Analog Scale (VAS) was applied before the intervention was performed, immediately after its implementation, and 24 hours later.
Pain reduction assessed by McGill Pain Scale | 24 hours
  The McGill Pain Scale was applied before the technique was performed and again after 24 hours.
Evaluate reduction of swelling using the REEDA scale. | 24 hours
  The REEDA scale was applied before the intervention was administered and again 24 hours after the intervention was performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT06370910/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT06370910/ICF_001.pdf